CLINICAL TRIAL: NCT05038319
Title: SAFETY AND EFFICACY OF ENDOSCOPIC CONVENTIONAL CYANOACRYLATE GLUE VS EUS-GUIDED COIL PLUS CYANOACRYLATE TECHNIQUE IN THE TREATMENT OF GASTRIC VARICES
Brief Title: SAFETY AND EFFICACY OF ENDOSCOPIC CONVENTIONAL CYANOACRYLATE GLUE VS EUS-GUIDED COIL PLUS CYANOACRYLATE TECHNIQUE IN THE TREATMENT OF GASTRIC VARICES: A RANDOMIZED CONTROLLED TRIAL
Acronym: GLUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, CLINICAL PROFESSOR, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUS GLUE 001
Record Dates: First submitted 2021-08-12; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Glue; Dependence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyanoacrylate injection and EUS guided coil and glue injection (Active Comparator): The procedure would be performed under conscious sedation.The endoscope would be used to reach the site of Varices. In Conventional technique treatment with cyanoacrylate the injection was performed using a 23-G sclerotherapy needle catheter . One vial of N-butyl-2-cyanoacrylate (0.5 mL) was mixed with Lipiodol) in a 1:1 ratio, and injected intravesically as a 1 mL bolus. The injection was repeated until total hardening of the varix. In treatment with coil and cyanoacrylate once the gastric varix was identified, the total diameter of the vascular pseudotumor was measured and the puncture was made at the site of the widest varix. The puncture was performed using a 19 G needle . the size of the coil after release should not be greater than the caliber of the vessel. Following coil deployment, 2 mL of distilled water was injected, followed by one vial (0.5 mL) of N-butyl-2-cyanoacrylate mixed with Lipiodol in 1:1 ratio.
  Interventions: Procedure: EUS
- COIL and GLUE (Placebo Comparator): Cyanoacrylate injection, first published by Soehendra in 1986, remains the conventional treatment method.
  Since coils were first used to treat ectopic varices by Levy in 2008(6), this technique has been increasingly implemented into clinical practice. However, its higher cost has been a limiting factor in more widespread use.
  Depending on the ectasia of the varix the following coil was deployed: 8 mm x 20 cm, 10 mm x 20 cm, or 10 mm x 30 cm (Interlock-18 Fibered IDC Occlusion System,Cook).
  Interventions: Procedure: EUS

INTERVENTIONS:
Procedure: EUS — The procedures would be performed by a therapeutic endoscope with the through the scope method. The endoscope would be used to reach the site of Varices.

SUMMARY:
To compare safety and efficacy of Endoscopic conventional technique (cyanoacrylate alone) to the EUS-guided injection technique (coil and cyanoacrylate) in the treatment of gastric varices.

Methods:

Patient recruitment:

Patients would be recruited from the endoscopy centre prior to their scheduled endoscopic intervention.

Study intervention :- Cyanoacrylate injection and EUS guided coil and glue injection The procedures would be performed by experienced endoscopists. The procedure would be performed under conscious sedation or monitored anaesthesia. The procedures would be performed by a therapeutic endoscope with the through the scope method. The endoscope would be used to reach the site of Varices. In Conventional technique treatment with cyanoacrylate the injection was performed using a 23-G sclerotherapy needle catheter (Interject®,Cook). One vial of N-butyl-2-cyanoacrylate (0.5 mL) was mixed with Lipiodol® in a 1:1 ratio, and injected intravesically as a 1 mL bolus. The injection was repeated until total hardening of the varix. In treatment with coil and cyanoacrylate once the gastric varix was identified, the total diameter of the vascular pseudotumor was measured and the puncture was made at the site of the widest varix. The puncture was performed using a 19 G needle (Expect®,Cook). The size of the coil used was selected based on the size of the widest varix in the pseudotumor; the size of the coil after release should not be greater than the caliber of the vessel. Following coil deployment, 2 mL of distilled water was injected, followed by one vial (0.5 mL) of N-butyl-2-cyanoacrylate mixed with Lipiodol in 1:1 ratio. Then, another 2 mL of distilled water was injected, and the needle was removed.

COIL and GLUE:

Cyanoacrylate injection remains the conventional treatment method. Since coils were first used to treat ectopic varices by Levy in 2008(6), this technique has been increasingly implemented into clinical practice. However, its higher cost has been a limiting factor in more widespread use.

Depending on the ectasia of the varix the following coil was deployed: 8 mm x 20 cm, 10 mm x 20 cm, or 10 mm x 30 cm (Interlock-18 Fibered IDC Occlusion System,Cook).

D.2.5 Randomization Patients were randomized into two groups: group I received standard endoscopic treatment with injection of a cyanoacrylate/Lipiodol (1:1) solution and group II received EUS-guided coiling and cyanoacrylate injection treatment A computer-based randomization list was generated with the online software Research Randomizer with 1:1 ratio (www.randomizer.org). An independent researcher not involved in this trial created the randomization list and sealed sequential opaque envelopes containing the random allocation sequence. The complete list generation occurred before the first enrollment.

D.2.6 Post-procedural management After the procedure, EUS with Doppler flow evaluation was repeated to check the presence or absence of flow within the varix. The patients remained under observation in the GI endoscopy unit for at least one hour, being released if no complaint was reported. After endoscopic treatment, all patients underwent thoracic and abdomen computerized tomography (CT) scanning within one week, independent of the development of clinical symptoms.

DETAILED DESCRIPTION:
All patients returned to the GI endoscopy unit approximately one month after initial endoscopic intervention for a repeat EUS evaluation.

Technical success is defined as complete obliteration of varices and absence of flow signal.On this occasion, if any residual flow was identified, new treatment was performed following the same technique initially used, and another evaluation was thus performed one month later. This scenario was repeated until complete thrombosis was achieved.

Complications that occurred during the procedure or within seven days post-intervention were defined as early complications, whereas those that occurred greater than or equal to seven days post-intervention were defined as late complications.

Recurrence was defined as evidence of any flow within the varix which occurred after initial obliteration had been confirmed.

5.Esophageal stricture 6.Iodine allergy (for EV)

Follow-up:

Once complete thrombosis was achieved, follow-up evaluations were performed three and nine months later (i.e. four and 10 months after therapy), at which time patients were questioned about any post-procedure complications, and underwent another EUS examination, which permitted repeat evaluations of flow within the treated vessel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, patients diagnosed with
* gastric varices larger than 2.0 cm in total diameter of the vascular pseudotumor type GOV2 or IGV 1.
* Active bleeder
* Secondary prophylaxis - h/o previous bleed
* High risk GV (GOV 2/IGV 1) - Baveno VI-
* Primary prophylaxis

Excusion criteria:

* Previous HRS
* MOF
* Platelet <50,000/cumm
* INR>2
* Esophageal stricture
* Iodine allergy (for EV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome was to compare the occurrence of embolism in the two groups | 4 months
  Technical success is defined as complete obliteration of varices and absence of flow signal.On this occasion, if any residual flow was identified, new treatment was performed following the same technique initially used, and another evaluation was thus performed one month later. This scenario was repeated until complete thrombosis was achieved.

SECONDARY OUTCOMES:
Secondary outcome was to evaluate the efficacy of the two techniques in the eradication of the varices. | 9 MONTHS
  Technical success is defined as complete obliteration of varices and absence of flow signal.On this occasion, if any residual flow was identified, new treatment was performed following the same technique initially used, and another evaluation was thus performed one month later. This scenario was repeated until complete thrombosis was achieved.

CONTACTS AND LOCATIONS:
Overall Officials: RAJESH GUPTA, MBBS MD, Study Director — ASIAN INSTITUTE OF GASTROENTEROLOGY PVT LTD
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India